CLINICAL TRIAL: NCT03518528
Title: Endometrial Estrogen Preparation Before Frozen-thawed Embryo Transfer : Comparison of Vaginal and Transdermal Administration
Brief Title: Comparison of Vaginal and Transdermal Oestrogen Before Frozen Thawed Embryo Transfer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PATCHS2018
Record Dates: First submitted 2018-03-24; First posted 2018-05-08 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-05

CONDITIONS: Embryo Transfer; Infertility
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transdermal: transdermal estradiol (Vivelledot, Novartis) 100 µg on day 3, then 200 µg day 7 and every 4 days, until first pregnancy test. If pregnancy test is positive, treatment is to continue until 8 weeks.
  Interventions: Drug: Estradiol 100 µg
- vaginal: Vaginal estradiol (Provames, Sanofi) 4mg per day from day 3 to first pregnancy test. If pregnancy test is positive, treatment is to continue until 8 weeks
  Interventions: Drug: Estradiol 2 MG

INTERVENTIONS:
Drug: Estradiol 2 MG — Vaginal estradiol (Provames, Sanofi) 4mg per day from day 3 to first pregnancy test. If pregnancy test is positive, treatment is to continue until 8 weeks
  Other Names: provames 2mg
  Groups: vaginal
Drug: Estradiol 100 µg — transdermal estradiol (Vivelledot, Novartis) 100 µg on day 3, then 200 µg day 7 and every 4 days, until first pregnancy test. If pregnancy test is positive, treatment is to continue until 8 weeks.
  Other Names: vivelledot 100 µg
  Groups: transdermal

SUMMARY:
The purpose of this study is to compare pregnancy outcomes of frozen-thawed embryo transfer after endometrial preparation with vaginal estradiol or transdermal estradiol and to evaluate women's satisfaction

DETAILED DESCRIPTION:
Frozen-thawed transfer embryo are more and more frequent but to date, there is no consensus on the ideal management of the adequate endometrial preparation.

Artificial preparation of endometrium is commonly used in assisted reproduction center because it is more easy to schedule.

Estradiol could be administrate by oral, vaginal or transdermal, but no protocol seems to improve clinical pregnancy rates.

To investigator's knowledge, transdermal estradiol has never been compare to vaginal administration before frozen-thawed embryo transfer.

Because transdermal administration could improve satisfaction of patients and reduce duration of treatment (when compare to oral administration), the investigators conduct a prospective study to compare clinical pregnancy rate after transdermal or vaginal estradiol administration to prepare the endometrium before frozen-thawed embryo transfer.

The investigator also evaluate side effects and patients satisfaction in both protocol.

The patients choose if they prefer vaginal or transdermal protocol after receiving sufficient information during medical consultation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and <43
* frozen-thawed embryo transfer after exogenously administered estrogen in either way transdermal or vaginal
* patients who accepted being included and signed the consent forms.

Exclusion Criteria:

* patient who refuse to participate
* frozen-thawed embryotransfer after stimulated or natural cycle
* oocyte or sperm donation
* endometrial thickness after 21 days <6mm
* non-french speaking patients
* women under legal guardianship
* women with no health or social security coverage

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: patients follow in our assisted reprodution unit, requesting frozen-thawed embryo transfer after ivf or icsi
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | 12 weeks
  defined as fetal cardiac activity at 12 weeks of gestation

SECONDARY OUTCOMES:
chemical pregnancy | 6 weeks
  Defined as serum HCG levels >10 IU/L, 14 days after the embryo transfer, followed by a rapid decrease until being undetectable
spontaneous pregnancy loss | 12 weeks
  Including early and late pregnancy losses
plasmatic estradiol concentration on the day of transfer | 21 days
  plasmatic estradiol concentration on the day of transfer
plasmatic lh concentration on the day of transfer | 21 days
  plasmatic lh concentration on the day of transfer
plasmatic progesterone concentration on the day of transfer | 21 days
  plasmatic progesterone concentration on the day of transfer
endometrial thickness | 21 days
  sonographic measurement of endometrial thickness on the day of transfer
annulation | 21 days
  defined when transfer is cancel if endometrial thickness is too thick (>6-7mm), when spontaneous ovulation is found with progesterone plasmatic increase and corpus luteum is seen by sonography or when unpredictable events occur (infections, ZIKA suspicion, endometriosis crisis, bad observance…). Annulation could be decided by biologist in case of embryo's lysis or bad quality seen after thawing.
treatment duration | 21 days
  duration of treatment before transfer
satisfaction evaluated by anonymous survey the day of transfer | 1 month
  evaluated by anonymous survey the day of transfer

CONTACTS AND LOCATIONS:
Overall Officials: BOUET Pierre Emmanuel, Study Director — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided